CLINICAL TRIAL: NCT03306420
Title: Phase I, First-in-Human, Open-Label, Multiple-Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Clinical Activity of MS201408-0005A as Single Agent and Sequentially in Combinations With MS201408-0005C or MS201408-0005B in Subjects With Metastatic or Locally Advanced Unresectable Solid Tumors
Brief Title: First-in-Human Study of MS201408-0005A as Single Agent and in Combinations
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated early due to lackluster pharmacodynamic data that showed no significant reduction of plasma kynurenine at steady state of M4112.
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS201408-0005
Record Dates: First submitted 2017-10-05; First posted 2017-10-11 (Actual); Results first posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-01

CONDITIONS: Metastatic or Locally Advanced Unresectable Solid Tumors
Keywords: MS201408-0005A; MS201408-0005B; MS201408-0005C; First-in-Human; Advanced solid tumors
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part IA Dose Escalation: M4112 100 mg (Experimental): Participants received an oral dose of 100 milligrams (mg) M4112 twice daily in 28-day cycles, starting from Day 1 of each cycle until confirmed disease progression or unacceptable toxicity (up to 15 Months).
  Interventions: Drug: M4112
- Part IA Dose Escalation: M4112 200 mg (Experimental): Participants received an oral dose of 200 mg M4112 twice daily in 28-day cycles, starting from Day 1 of each cycle until confirmed disease progression or unacceptable toxicity (up to 15 Months).
  Interventions: Drug: M4112
- Part IA Dose Escalation: M4112 400 mg (Experimental): Participants received an oral dose of 400 mg M4112 twice daily in 28-day cycles, starting from Day 1 of each cycle until confirmed disease progression or unacceptable toxicity (up to 15 Months).
  Interventions: Drug: M4112
- Part IA Dose Escalation: M4112 600 mg (Experimental): Participants received an oral dose of 600 mg M4112 twice daily in 28-day cycles, starting from Day 1 of each cycle until confirmed disease progression or unacceptable toxicity (up to 15 Months).
  Interventions: Drug: M4112
- Part IA Dose Escalation: M4112 800 mg (Experimental): Participants received an oral dose of 800 mg M4112 twice daily in 28-day cycles, starting from Day 1 of each cycle until confirmed disease progression or unacceptable toxicity (up to 15 Months).
  Interventions: Drug: M4112

INTERVENTIONS:
Drug: M4112 — All participants who received M4112 100,200,400,600 and 800 mg twice daily in 28-day cycles, starting from Day 1 of each cycle until confirmed disease progression or unacceptable toxicity (up to 15 Months).

SUMMARY:
This is a Phase I, open-label study to determine the safety, tolerability, pharmacokinetic (PK), pharmacodynamics (PD), and preliminary antitumor activity of MS201408-0005A as single agent (Part IA only) and in combination with MS201408-0005C or MS201408-0005B (Part IB, Part IC).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with histologically or cytologically proven advanced or metastatic solid malignancies for whom no effective standard therapy exists or has failed or subjects who are intolerant to established therapy known to provide clinical benefit for their condition (dose escalation cohorts; Part I).
* An eastern cooperative oncology group performance status (ECOG PS) of 0 to 1 at screening and adequate hematological, renal and hepatic function as defined by protocol specified criteria.
* Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

* Intolerance to immune checkpoint inhibitor therapy as defined by the occurrence of an adverse drug reaction requiring drug discontinuation (dose escalation cohorts), concurrent anticancer treatment or immunosuppressive agents.
* Prior organ transplantation including allogeneic stem cell transplantation, brain metastases (except those meeting certain protocol specified criteria which are acceptable), significant acute or chronic infections, a history of cardiovascular/cerebrovascular disease.
* Current significant cardiac conduction abnormalities and hypokalemia as specified in the protocol.
* Warfarin or other Vitamin K antagonists treatment, strong inhibitors or inducers of cytochrome P450 (CYP)3A4, and drugs with a narrow therapeutic index, which are predominantly metabolized by CYP3A4 and drugs known to have a high risk to prolong QTc as per label.
* Pregnancy or lactation.
* Severe hypersensitivity reactions to monoclonal antibodies, known hypersensitivity to the investigational medicinal products or to one or more of the excipients, autoimmune diseases (inflammatory bowel diseases, interstitial lung disease, or pulmonary fibrosis), and live vaccines within 28 days prior to study entry.
* Pneumonitis and history of pneumonitis.
* Other protocol defined exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Inc., a business of Merck KGaA, Darmstadt, Germany
Locations (3):
- United States (3):
  - Yale Cancer Center, New Haven, Connecticut
  - University of TX M.D. Anderson Cancer Center-Investigational Cancer Therapeutics Partner, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas

REFERENCES:
- [Derived] Naing A, Eder JP, Piha-Paul SA, Gimmi C, Hussey E, Zhang S, Hildebrand V, Hosagrahara V, Habermehl C, Moisan J, Papadopoulos KP. Preclinical investigations and a first-in-human phase I trial of M4112, the first dual inhibitor of indoleamine 2,3-dioxygenase 1 and tryptophan 2,3-dioxygenase 2, in patients with advanced solid tumors. J Immunother Cancer. 2020 Aug;8(2):e000870. doi: 10.1136/jitc-2020-000870. PMID 32843490

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Participant First Visit: 03-Oct-2017 Last Participant Last Visit: 14-Jan-2019.
Groups:
- Part 1A Dose Escalation: M4112 100 mg: Participants received an oral dose of 100 milligrams (mg) M4112 twice daily in 28-day cycles, starting from Day 1 of each cycle until confirmed disease progression or unacceptable toxicity (up to 15 Months).
- Part 1A Dose Escalation: M4112 200 mg: Participants received an oral dose of 200 mg M4112 twice daily in 28-day cycles, starting from Day 1 of each cycle until confirmed disease progression or unacceptable toxicity (up to 15 Months).
- Part 1A Dose Escalation: M4112 400 mg: Participants received an oral dose of 400 mg M4112 twice daily in 28-day cycles, starting from Day 1 of each cycle until confirmed disease progression or unacceptable toxicity (up to 15 Months).
- Part 1A Dose Escalation: M4112 600 mg: Participants received an oral dose of 600 mg M4112 twice daily in 28-day cycles, starting from Day 1 of each cycle until confirmed disease progression or unacceptable toxicity (up to 15 Months).
- Part 1A Dose Escalation: M4112 800 mg: Participants received an oral dose of 800 mg M4112 twice daily in 28-day cycles, starting from Day 1 of each cycle until confirmed disease progression or unacceptable toxicity (up to 15 Months).
Period: Overall Study
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Started | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.7 (14.84) | 54.7 (8.33) | 43.0 (9.54) | 67.7 (7.51) | 62.3 (14.84) | 57.7 (13.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 3 | 3 | 13
  Male | 1 | 0 | 1 | 0 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 1 | 0 | 3
  Not Hispanic or Latino | 2 | 3 | 2 | 2 | 3 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 1 | 3
  White | 2 | 3 | 2 | 3 | 2 | 12
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1A Dose Escalation: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs) as Per National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03
Description: DLTs was assessed as per NCI CTCAE v 4.03. DLT defined as any Grade greater than or equal (>=) 3 nonhematological AE or Immune-related adverse event (irAE) assessed by Investigator or Sponsor during first Cycle (first 28 days) of study treatment. Asymptomatic Grade >= 3 lipase or amylase elevation not associated with clinical manifestations of pancreatitis. Any TEAE observed in subsequent cycle. Any Grade 4 neutropenia of >= 5 days duration, Grade >= 3 febrile neutropenia, Grade 3 hemoglobin decrease despite blood transfusion or erythroid growth factor. Grade 4 hemoglobin decrease assessed as related to study drug. Any Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with bleeding. Any Grade >= 3 clinical signs and symptoms related to increased QTc.
Time Frame: Cycle 1 (Each Cycle is of 28 days)
Population: DLT analysis set included all participants treated in dose escalation cohorts who do not miss greater than (>) 5 planned total daily doses of M4112 in the first cycle (first 28 days) of the dose escalation part for other than DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
Participants | 0 | 0 | 0 | 0 | 1

2. Primary Outcome: Part 1A Dose Escalation: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Who Experienced a Treatment Related Adverse Events (TRAE) According to National Cancer Institute Common Toxicity Criteria for Adverse Events Version 4.03
Description: An adverse event (AE) was defined as any untoward medical occurrence in participant which does not necessarily have casual relationship with treatment was any unfavorable and unintended sign(including abnormal laboratory finding), symptom/disease temporally associated with use of medicinal product, whether/not considered related to medicinal product. A serious adverse event(SAE) was AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Term TEAE is defined as AEs starting/worsening after first intake of the study drug. TEAEs included both Serious TEAEs and non-serious TEAEs. Treatment related AE was defined as having a "Possible" or "Related" relationship to study treatment, as assessed by the Investigator.
Time Frame: Baseline up to safety follow-up visit, assessed up to 15.4 months
Population: The safety analysis set included all participants who had received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
Participants
  Any TEAE | 3 | 3 | 3 | 3 | 3
  Any Related TEAE | 3 | 2 | 1 | 3 | 3

3. Primary Outcome: Part 1A Dose Escalation: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters
Description: The laboratory measurements included hematology, biochemistry and hormonal tests. Number of participants with any clinically significant abnormalities in laboratory measurements were reported. Clinical significance was determined by the investigator.
Time Frame: Baseline up to safety follow-up visit, assessed up to 15.4 months
Population: The safety analysis set included all participants who had received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
Participants | 1 | 0 | 0 | 0 | 1

4. Primary Outcome: Part 1A Dose Escalation: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Vital signs assessment included blood pressure, pulse rate and body temperature. Number of Participants with any clinically significant abnormalities in vital signs were reported. Clinical significance was determined by the investigator.
Time Frame: Baseline up to safety follow-up visit, assessed up to 15.4 months
Population: The safety analysis set included all participants who had received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
Participants | 2 | 0 | 1 | 1 | 1

5. Primary Outcome: Part 1A Dose Escalation: Number of Participants With On-Treatment Shift in Eastern Cooperative Oncology Performance Status (ECOG PS) Score From 0 to 1
Description: ECOG PS score is widely used by doctors and researchers to assess how a participants' disease is progressing, and is used to assess how the disease affects the daily living abilities of the participant, and determine appropriate treatment and prognosis. The score ranges from Grade 0 to Grade 4, where Grade 0 = Fully active, able to carry on all pre-disease performance without restriction, Grade 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (like light house work, office work), Grade 2 = Ambulatory and capable of all self-care but unable to carry out any work activities, Grade 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours and Grade 4 = Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair. Number of participants with on-treatment shift in ECOG PS Score from 0 to 1 were reported.
Time Frame: Baseline up to safety follow-up visit, assessed up to 15.4 months
Population: The safety analysis set included all participants who had received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
Participants | 1 | 0 | 1 | 0 | 1

6. Primary Outcome: Part 1A Dose Escalation: Number of Participants With Clinically Significant Change From Baseline in Physical Examination Abnormalities
Description: A complete physical examination (including, general appearance, skin, pulmonary, cardiovascular, gastrointestinal, external genitourinary only as medically relevant, lymphatic, neurologic and musculoskeletal systems, head/neck, extremities, eyes, ears, nose, throat, and cognitive status) was performed. Number of participants with clinical significant change from baseline in physical examination abnormalities were reported. Clinical significance was determined by the investigator.
Time Frame: Baseline up to safety follow-up visit, assessed up to 15.4 months
Population: The safety analysis set included all participants who had received at least 1 dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Part 1A Dose Escalation: Area Under the Plasma Concentration Curve From Time Zero to 8 Hours Post Dose AUC(0-8h) of M4112
Description: Area under the drug concentration-time curve from 0 to 8 h post dosing for M4112. AUC0-8 was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6 and 8 h post-dose on Day 1 and 15 of Cycle 1 (Each Cycle is for 28 days)
Population: Pharmacokinetic (PK) analysis set included all participants who received M4112 and for whom at least 1 dose of M4112 and must have sufficient M4112 plasma concentration data to enable the calculation of at least 1 PK parameter. Here "number analyzed" signifies those participants who were evaluable for this outcome measure at given time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
nanogram*hour per milliliter (ng*h/mL)
  Cycle 1 Day 1 | 3550 (14.4) | 8740 (13.6) | 27700 (21.4) | 50400 (7.7) | 14600 (85.1)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1
  Cycle 1 Day 15 | 4790 (25.4) | 7580 (11.5) | 31500 (28.8) | 59500 (12.7) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated as it was pre-specified not to calculate the Descriptive statistics if less than 3 number of participants. Individual value was 93200 ng*h/mL.

8. Secondary Outcome: Part 1A Dose Escalation: Maximum Observed Plasma Concentration (Cmax) of M4112
Description: Pharmacokinetic PK parameter Cmax was obtained directly from the plasma concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6 and 8 h post-dose on Day 1 and 15 of Cycle 1 (Each Cycle is for 28 days)
Population: PK analysis set included all participants who received M4112 and for whom at least 1 dose of M4112 and must have sufficient M4112 plasma concentration data to enable the calculation of at least 1 PK parameter. Here "number analyzed" signifies those participants who were evaluable for this outcome measure at given time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 | 806 (9.9) | 2110 (13.6) | 7670 (39.6) | 11700 (24.6) | 2770 (83.6)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1
  Cycle 1 Day 15 | 975 (34.9) | 1720 (20.5) | 6560 (27.4) | 12100 (2.2) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated as it was pre-specified not to calculate the Descriptive statistics if less than 3 number of participants. Individual value was 21100 ng/mL.

9. Secondary Outcome: Part 1A Dose Escalation: Time to Reach Maximum Plasma Concentration (Tmax) of M4112
Description: Time to reach the maximum plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6 and 8 h post-dose on Day 1 and 15 of Cycle 1 (Each Cycle is for 28 days)
Population: as for outcome 8
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
Hours
  Cycle 1 Day 1 | 1.08 [1.08 to 2.12] | 2.10 [2.07 to 3.08] | 1.08 [1.07 to 1.08] | 1.00 [0.97 to 1.07] | 2.08 [2.07 to 4.12]
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1
  Cycle 1 Day 15 | 3.08 [2.12 to 4.13] | 2.10 [1.00 to 6.08] | 1.08 [0.50 to 3.00] | 1.03 [0.93 to 2.17] | NA [2.00 to 2.00] — Median was not calculated as it was pre-specified not to calculate the Descriptive statistics if less than 3 number of participants. Individual value was 2.00 hours.

10. Secondary Outcome: Part 1A Dose Escalation: Dose Normalized Area Under the Plasma Concentration-Time Curve From Time Zero to 8 Hour Post-dose (AUC0-8/Dose) of M4112
Description: Dose normalized was calculated as area under the plasma concentration-time curve from time zero to 8 h postdose divided by dose.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6 and 8 h post-dose on Day 1 and 15 of Cycle 1 (Each Cycle is for 28 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
ng*h/mL/mg
  Cycle 1 Day 1 | 35.5 (14.4) | 43.7 (13.6) | 69.1 (21.4) | 84.0 (7.7) | 18.2 (85.1)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1
  Cycle 1 Day 15 | 47.9 (25.4) | 37.9 (11.5) | 78.8 (28.8) | 99.2 (12.7) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated as it was pre-specified not to calculate the Descriptive statistics if less than 3 number of participants. Individual value was 116 ng*h/mL/mg.

11. Secondary Outcome: Part 1A Dose Escalation: Dose Normalized Maximum Observed Plasma Concentration (Cmax/Dose) of M4112
Description: Dose normalized was calculated as Cmax obtained directly from the concentration versus time curve divided by dose.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6 and 8 h post-dose on Day 1 and 15 of Cycle 1 (Each Cycle is for 28 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
ng/mL/mg
  Cycle 1 Day 1 | 8.06 (9.9) | 10.5 (13.6) | 19.2 (39.6) | 19.6 (24.6) | 3.47 (83.6)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1
  Cycle 1 Day 15 | 9.75 (34.9) | 8.58 (20.5) | 16.4 (27.4) | 20.2 (2.2) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated as it was pre-specified not to calculate the Descriptive statistics if less than 3 number of participants. Individual value was 26.4 ng/mL/mg.

12. Secondary Outcome: Part 1A Dose Escalation: Accumulation Ratio for Area Under the Plasma Concentration-Time Curve From Time Zero to 8 Hour Post-dose (Racc[AUC0-8h]) of M4112
Description: Accumulation ratio for Area Under the Plasma Concentration-Time Curve From Time Zero to 8 hours After Administration (Racc[AUC0-8h]) of M4112 was reported. Racc(AUC0-8h) calculated as AUC0-8h, on Cycle 1 Day 15 divided by AUC0-8h on Cycle 1 Day 1.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6 and 8 h post-dose on Day 1 and 15 of Cycle 1 (Each Cycle is for 28 days)
Population: PK analysis set included all participants who received M4112 and for whom at least 1 dose of M4112 and must have sufficient M4112 plasma concentration data to enable the calculation of at least 1 PK parameter. Here "Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 1
Ratio | 1.35 (11.4) | 0.868 (15.3) | 1.14 (50.1) | 1.18 (9.4) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated as it was pre-specified not to calculate the Descriptive statistics if less than 3 number of participants. Individual value was 4.67.

13. Secondary Outcome: Part IA Dose Escalation: Accumulation Ratio for Maximum Observed Plasma Concentration (Racc [Cmax]) of M4112
Description: Accumulation ratio for Cmax was calculated as Cmax, Cycle 1 Day 15 divided by Cmax, Cycle 1 Day 1.
Time Frame: Pre-dose, 0.5, 1, 2, 3, 4, 6 and 8 h post-dose on Day 1 and 15 of Cycle 1 (Each Cycle is for 28 days)
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 1
Ratio | 1.21 (24.8) | 0.815 (7.0) | 0.856 (66.8) | 1.03 (23.0) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated as it was pre-specified not to calculate the Descriptive statistics if less than 3 number of participants Individual value was 5.26.

14. Secondary Outcome: Part 1A Dose Escalation: Pre-dose Observed Plasma Concentration (Cpre) of M4112
Description: Maximum pre-dose observed plasma concentration was reported.
Time Frame: Pre-dose on Days 8, 15 (Cycle 1) and Day 1 (Cycle 2) (Each Cycle is 28 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
ng/mL
  Cycle 1 Day 8 | 156 (58.2) | 96.5 (85.0) | 1240 (51.6) | 4410 (54.5) | 5200 (105.4)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1
  Cycle 1 Day 15 | 221 (20.5) | 199 (53.9) | 1630 (45.7) | 3380 (42.4) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated as it was pre-specified not to calculate the Descriptive statistics if less than 3 number of participants. Individual value was 9810 ng/mL.
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 2 | 3 | 2 | 1
  Cycle 2 Day 1 | 128 (67.7) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated as it was pre-specified not to calculate the Descriptive statistics if less than 3 number of participants. Individual values were 83.3 and 85.2 ng/mL. | 957 (72.1) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated as it was pre-specified not to calculate the Descriptive statistics if less than 3 number of participants. Individual values were 1910 and 2560 ng/mL. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated as it was pre-specified not to calculate the Descriptive statistics if less than 3 number of participants. Individual value was 8560 ng/mL.

15. Secondary Outcome: Part 1A Dose Escalation: Dose Normalized Pre-dose Observed Plasma Concentration (Cpre/Dose) of M4112
Description: Dose normalized pre-dose observed plasma concentration (Cpre/dose) of M4112 was reported.
Time Frame: Pre-dose on Days 8, 15 (Cycle 1) and Day 1 (Cycle 2) (Each Cycle is 28 days)
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
ng/mL/mg
  Cycle 1 Day 8 | 1.56 (58.2) | 0.482 (85.0) | 3.11 (51.6) | 7.35 (54.5) | 6.50 (105.4)
  Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 3 | 3 | 1
  Cycle 1 Day 15 | 2.21 (20.5) | 0.997 (53.9) | 4.08 (45.7) | 5.63 (42.4) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated as it was pre-specified not to calculate the Descriptive statistics if less than 3 number of participants. Individual value was 12.3 ng/mL/mg.
  Cycle 2 Day 1: number analyzed (Participants) | 3 | 2 | 3 | 2 | 1
  Cycle 2 Day 1 | 1.28 (67.7) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated as it was pre-specified not to calculate the Descriptive statistics if less than 3 number of participants. Individual values were 0.417 and 0.426 ng/mL/mg. | 2.39 (72.1) | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated as it was pre-specified not to calculate the Descriptive statistics if less than 3 number of participants. Individual values were 3.18 and 4.27 ng/mL/mg. | NA (NA) — Geometric Mean and Geometric Coefficient of Variation were not calculated as it was pre-specified not to calculate the Descriptive statistics if less than 3 number of participants. Individual value was 10.7 ng/mL/mg.

16. Secondary Outcome: Part 1A Dose Escalation: Slope of Concentration-QTc (cQTc) Regression of M4112
Description: Time-matched, replicate ECGs and PK samples collected in the dose-escalation phase and planned to analyze QTC response using slope analysis of exposure/response.
Time Frame: Baseline up to safety follow-up visit, assessed up to 15.4 months
Population: Data was not collected as the study was prematurely terminated due to lackluster pharmacodynamic data.
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Part 1A Dose Escalation: Number of Participants With Best Overall Response (BOR)
Description: BOR was determined according to Response Evaluation Criteria in Solid Tumors version1.1(RECIST 1.1).Best response obtained among all tumor assessment visits after the date of first study drug administration until documented disease progression. BOR rate is defined as the number of participants with BOR was either confirmed complete response (CR) partial response (PR), stable disease (SD) and progressive disease (PD) relative to the number of participants belonging to the study of interest. CR:Disappearance of all target lesions; PR:At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD; PD:At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; SD:Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: From first dose of study drug administration until PD, assessed up to 15.4 months
Population: The safety analysis set included all participants who had received at least 1 dose of the study treatment. Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 2
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0
  Stable Disease | 2 | 3 | 3 | 1 | 0
  Progressive Disease | 1 | 0 | 0 | 2 | 2

18. Secondary Outcome: Part 1A Dose Escalation: Duration of Response
Description: Duration of response defined as time from first documentation of objective response complete response (CR) or partial response (PR) whichever is first recorded) to date of first documentation of objective progression of disease or death due to any cause whichever occurs first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of longest diameter (SLD) of all lesions.
Time Frame: From first dose of study drug administration until PD, assessed up to 15.4 months
Population: Data was not collected as the study was prematurely terminated due to lackluster pharmacodynamic data.
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Part 1A Dose Escalation: Disease Control Rate
Description: Disease control was defined as percentage of participants with complete response (CR), partial response (PR), or stable disease (SD) as the best overall response according to radiological assessments as adjudicated by the IRC from randomization until the first occurrence of PD. CR defined as disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR defined as at least a 30% decrease in the sum of diameters of target lesions taking as reference the baseline sum diameters. PD was defined as an increase of at least 20% in the sum of the diameters of target lesions, taking as reference the smallest sum of the diameters of target lesions recorded since treatment started. Percentage of participants with disease control were reported.
Time Frame: From first dose of study drug administration until PD, assessed up to 15.4 months
Population: The safety analysis set included all participants who had received at least 1 dose of the study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
Percentage of Participants | 66.7 [9.4 to 99.2] | 100 [29.2 to 100.0] | 100 [29.2 to 100.0] | 33.3 [0.8 to 90.6] | 0.0 [0.0 to 70.8]

20. Secondary Outcome: Part 1A Dose Escalation: Time to Tumor Response
Description: Tumor response was defined as the presence of at least 1 confirmed complete response (CR) or confirmed partial response (PR) as judged by RECIST version 1.1. CR was defined for target lesions (TLs) as the disappearance of all lesions, and for non-target lesions (NTLs) as the disappearance of all non-target non-measurable lesions and/or normalization of serum levels of tumor markers. PR was defined for TLs as at least a 30 percent (%) decrease from baseline (BL) in the sum of longest diameter (SLD) of TLs.
Time Frame: From first dose of study drug administration until PD, assessed up to 15.4 months
Population: Data was not collected as the study was prematurely terminated due to lackluster pharmacodynamic data.
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Part 1A Dose Escalation: Progression Free Survival Time (PFS)
Description: Progression free survival time defined as time from start date to the date of the first documentation of objective progression of disease or death due to any cause, whichever occurs first. PD was defined as at least a 20 percent (%) increase in the sum of longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. PFS was measured using Kaplan-Meier (KM) estimates.
Time Frame: From first dose of study drug administration until PD, assessed up to 15.4 months
Population: The safety analysis set included all participants who had received at least 1 dose of the study treatment.
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3
Months | 3.7 [1.9 to 8.1] | 5.5 [3.9 to 5.5] | NA [2.1 to 10.2] — The Median was not reached due to higher number (>50%) of censored participants. | 1.8 [1.1 to 3.7] | 1.2 [0.0 to 1.2]

ADVERSE EVENTS:
Time Frame: Baseline up to safety follow-up visit, assessed up to 15.4 months
Arm/Group | Part 1A Dose Escalation: M4112 100 mg | Part 1A Dose Escalation: M4112 200 mg | Part 1A Dose Escalation: M4112 400 mg | Part 1A Dose Escalation: M4112 600 mg | Part 1A Dose Escalation: M4112 800 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/3 | 1/3 | 1/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A Dose Escalation: M4112 100 mg (N=3) | Part 1A Dose Escalation: M4112 200 mg (N=3) | Part 1A Dose Escalation: M4112 400 mg (N=3) | Part 1A Dose Escalation: M4112 600 mg (N=3) | Part 1A Dose Escalation: M4112 800 mg (N=3)
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A Dose Escalation: M4112 100 mg (N=3) | Part 1A Dose Escalation: M4112 200 mg (N=3) | Part 1A Dose Escalation: M4112 400 mg (N=3) | Part 1A Dose Escalation: M4112 600 mg (N=3) | Part 1A Dose Escalation: M4112 800 mg (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 0 | 1 | 1 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Amylase increased (Investigations) | 0 | 0 | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1 | 1
Blood urea increased (Investigations) | 0 | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1
Lipase increased (Investigations) | 0 | 1 | 0 | 2 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Part IB and Part IC for this study were never initiated as the study was terminated early due to lackluster pharmacodynamic data that showed no significant reduction of plasma kynurenine at steady state at a range of tested dose levels of M4112.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT03306420/SAP_000.pdf
  • Study Protocol (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT03306420/Prot_001.pdf